CLINICAL TRIAL: NCT03265392
Title: Digestion: Building a Better Health and Better Understanding the Digestive Processes Thanks to Magnetic Resonance Imaging
Brief Title: Impact of Food Combination on Starch Digestion and Gastric Processing
Acronym: DECOUVRIR-M
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: IR4M (Imagerie par Résonance Magnétique Médicale et Multi-Modalités) (Unknown)
Responsible Party: Principal Investigator, Robert Benamouzig, Professor, MD, PhD, Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: DECOUVRIR-M
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Glycemic Index; Gastric Emptying; Appetite
MeSH Terms: interventions — Bread; Water; Tea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part 1 - Bread + Water (Other): Participants in this arm will randomly consume bread and 250 mL of water on 1 out of 3 visits of Part 1.
  Interventions: Other: Bread; Other: Water
- Part 1 - Bread + Lemon Juice (Other): Participants in this arm will randomly consume bread and 250 mL of lemon juice on 1 out of 3 visits of Part 1.
  Interventions: Other: Bread; Other: Lemon juice
- Part 1 - Bread + Tea (Other): Participants in this arm will randomly consume bread and 250 mL of tea on 1 out of 3 visits of Part 1.
  Interventions: Other: Bread; Other: Tea
- Part 2 - Bread + water (Other): Participants in this arm will randomly consume bread and 250 mL of water supplemented with 20 peas on 1 out of 3 visits of Part 2.
  Interventions: Other: Bread; Other: Water; Other: Peas
- Part 2 - Bread+ Lemon Juice (Other): Participants in this arm will randomly consume bread and 250 mL of lemon juice supplemented with 20 peas on 1 out of 3 visits of Part 2.
  Interventions: Other: Bread; Other: Lemon juice; Other: Peas
- Part 2 - Bread+ tea (Other): Participants in this arm will randomly consume bread and 250 mL of tea supplemented with 20 peas on 1 out of 3 visits of Part 2.
  Interventions: Other: Bread; Other: Tea; Other: Peas

INTERVENTIONS:
Other: Bread — Serving of wheat bread providing 50 g of carbohydrates
Other: Water — 250 mL of water
  Arms: Part 1 - Bread + Water; Part 2 - Bread + water
Other: Lemon juice — 250 mL of lemon juice
  Arms: Part 1 - Bread + Lemon Juice; Part 2 - Bread+ Lemon Juice
Other: Tea — 250 mL of tea
  Arms: Part 1 - Bread + Tea; Part 2 - Bread+ tea
Other: Peas — 20 peas
  Arms: Part 2 - Bread + water; Part 2 - Bread+ Lemon Juice; Part 2 - Bread+ tea

SUMMARY:
The results of our in vitro studies strengthen the hypothesis that the contribution of salivary alpha-amylase to starch digestion has been underrated and that this enzyme can play an important role in this process. As a result, its inhibition could constitute an opportunity to reduce the glycemic response elicited by starch-rich foods. The main goal of this study is to verify whether inhibiting salivary alpha-amylase upon the consumption of starchy foods, can have an impact on the postprandial glycemic response, and/or satiety.

DETAILED DESCRIPTION:
The main objective of this work was to test the impact of adding black tea or lemon juice to a starch-rich meal on postprandial plasma glucose concentrations and on energy intake in healthy humans. This study was divided into two parts.

The objective of part 1 was to determine the effect of pairing a starch-rich food with water, black tea or lemon juice on postprandial plasma glucose and energy intake in healthy humans. This study was conducted in semi-controlled conditions. The three test meals (equal portions of bread (100 g) and 250 mL of either water, black tea or lemon juice) were consumed as breakfast (after a 10-h fast) on independent days and in a randomised order. Capillary blood glucose concentrations were self-monitored using the finger-prick method at pre-defined time-points during 180 min. Ad libitum energy intake was assessed 3 hours later.

The main objective of part 2 was to investigate whether the gastric emptying patterns remain, or not, the same when a bread meal is paired with water, tea, and lemon juice. Blood glucose response and satiety perceptions were also monitored. The test meals were similar to those in branch 1, except that the meals were supplemented with 20 peas, which the subjects were asked to swallow at the end (with half of the beverage provided) without chewing. These peas conferred a distinct contrast in MRI scans and could be used as stomach motility and gastric mixing tracers in MRI images. Capillary blood glucose concentrations were determined using the finger-prick method at pre-defined time-points during 180 min. Visual analogue scales were used to assess satiety-related perceptions.

Volunteer recruitment was conducted independently for each part of the study and volunteers were allowed to participate in one part of the study only. Data collected in each part of the study was analysed independently.

ELIGIBILITY:
Inclusion Criteria:

* To be overall healthy
* To be between 18 and 60 years old
* BMI between 18 and 25 (lean)
* No eating disorders
* No major weight changes (> 3kg in previous 3 months)
* Structured eating habits (3 main meals/day, everyday)
* Not using corticoid drugs, or antidepressives known to influence food consumption, appetite and/or mood.
* Not using medication known to influence glucose tolerance: acetylsalicylic acid or thyroxin, vitamin or mineral-based dietary supplements, and drugs to control hypertension or osteoporosis are acceptable
* No allergies to the foods in the test-meals and ad libitum meal
* No abusive alcohol consumption
* No intensive exercising habits
* No participation in a clinical study within the previous 6 months
* To enjoy the foods in the test-meals and ad libitum meals
* To be affiliated to a social security system
* To be available to participate in study sessions
* To have read and signed the Informed consent form

Additional criteria for Part 2

* Male
* Ability to be in an MRI scan without moving
* Ability to hold breath for 25s (a requirement for certain MRI exams)

Non-inclusion criteria:

* History of diabetes, use of antihyperglycemic drugs or insulin to treat diabetes or associated conditions
* Major medical interventions or surgeries requiring hospitalization within the previous 3 months
* Any medical condition that affects digestion and/or nutrient absorption
* Use of steroids, protease inhibitors and/or antipsychotic drugs
* Use of anticoagulation drugs
* To be participating in another clinical trial, or to be within the exclusion period of a previous clinical trial
* To have started or stopped smoking within the previous 3 months

Additional exclusion criteria for Part 2:

* Any contraindications to an MRI exam: claustrophobia, tatoos, presence of ferromagnetic elements, having a pacemaker, metallic prosthesis, cochlear implants, vascular clips, insulin pumps
* Any condition or disease that might affect the results of MRI exams.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2018-07-06 (Actual); Study Completion 2018-07-06 (Actual)

PRIMARY OUTCOMES:
Energy intake (Main outcome of Part 1) | 3 hours
  Consumption at an ad libitum meal served 3 h after each test-meal during part 1
Gastric emptying (Main outcome of Part 2) | 3 hours
  Gastric empting kinetics of each test-meal, evaluated by MRI, during part 2

SECONDARY OUTCOMES:
Glycemic Response (Secondary outcome of Parts 1 and 2) | At baseline and and at different time-points during 3 hours after after consuming the test meal
  Capillary blood glucose monitoring
Subjective appetite sensations (Secondary outcome of Part 2) | At baseline and at different time-points during 3 hours after consuming the test meal
  Evaluation of satiety, fullness, hunger, prospective food consumption and desire to eat through visual analogue scales (VAS)

OTHER OUTCOMES:
End of the day questionnaire | 12-16 hours after the test meal (Part 1 and 2)
  Digital questionnaire that will be answered at the end of the day in order to provide a reference point regarding the potential effects of the test-meal throughout the rest of the day (ex. appetite, food consumption, discomfort sensations)
Gastric contractions | At baseline and during 3 hours after after consuming the test meal (Part 2 only)
  Analysis of MRI scans will be carried out to evaluate the frequency of gastric contractions.
Amylolytic activity of saliva | At baseline (Part 1)
  The amylolytic activity of saliva samples collected before the test meal will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Benamouzig, MD, PhD, Principal Investigator — Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Locations (1):
- Centre de Recherche sur Volontaires (CRV), Hospital Avicenne, Bobigny, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Freitas D, Boue F, Benallaoua M, Airinei G, Benamouzig R, Lutton E, Jourdain L, Dubuisson RM, Maitre X, Darrasse L, Le Feunteun S. Glycemic response, satiety, gastric secretions and emptying after bread consumption with water, tea or lemon juice: a randomized crossover intervention using MRI. Eur J Nutr. 2022 Apr;61(3):1621-1636. doi: 10.1007/s00394-021-02762-2. Epub 2022 Jan 11. PMID 35013789